CLINICAL TRIAL: NCT05647148
Title: The Effect of Progressive Relaxation Exercises on Sleep Quality, Serotonin, and Melatonin Levels of Heart Diseases Patients
Brief Title: The Effect of Progressive Relaxation Exercises on Sleep Quality
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Tunc ELIS, LECTURER, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AU-TELIS
Record Dates: First submitted 2022-11-21; First posted 2022-12-12 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Sleep Disturbance; Nursing Care
Keywords: sleep quality; progressive relaxation Exercises; melatonin; serotonin
MeSH Terms: conditions — Parasomnias; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: randomized controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): progressive relaxiation exercises Will do sixty minutes of progressive relaxation exercise for three consecutive days
  Interventions: Behavioral: Progressive Relaxation Exercises
- Control group: (No Intervention): no intervention

INTERVENTIONS:
Behavioral: Progressive Relaxation Exercises — In the first part of this audio material, which consists of three parts; The definition of deep relaxation, its purpose and points to be considered during exercise are included.
  The second part, consisting of an average of thirty minutes, includes the explanation of relaxation exercises with verbal commands accompanied by the sound of the stream.
  In the last part, there is only relaxation music without any commands.
  Arms: intervention group

SUMMARY:
This study; In order to investigate the effect of progressive relaxation exercises on sleep quality, serotonin and melatonin levels in cardiac patients with sleep problems, a pretest/posttest experimental design study will be conducted with a control group.

The data of this study will be collected between May 2022 and December 2022. The research will be carried out with a total of 60 (experimental group=30, control group=30) patients treated for heart failure, myocardial infarction and angina pectoris in the cardiology clinic of a university hospital.

The data of the study will be collected using the Richard's Campbell Sleep Scale and the Commercial ELISA kit.

Progressive relaxation exercises will be applied to the patients included in the experimental group for 3 consecutive days.

Before relaxation exercises, urine melatonin, serotonin level [5-hydroxyindolacetic acid (5-HIAA) and 6-sulphatoxymelatonin(6-HMS)] measurement and sleep quality will be measured according to the kit procedure.

In the analysis of the data, significance p <0.05 will be accepted. Institutional permission, ethics committee approval, and written consent from the participants were obtained before the study.

DETAILED DESCRIPTION:
The data of this study will be collected between May 2022 and December 2022. The research will be carried out with a total of 60 (experimental group=30, control group=30) patients treated for heart failure, myocardial infarction and angina pectoris in the cardiology clinic of a university hospital.

The study was planned as a randomized controlled experiment. Patients meeting the research criteria will be randomly assigned to 30 experimental-30 control groups by randomization method.

Information Form, Richard's Campbell Sleep Scale and commercial ELISA kit will be used as data collection tools in the research.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years of age,
* who reported sleep problems
* scored 25 or less on the Richard's Campbell Sleep Scale,
* were scheduled to be hospitalized for at least 4 days,
* had no pain, were able to give urine samples,
* were lying in a single or double room,
* had serotonin-containing or decreased serotonin secretion.
* do not take any medication that provides medical treatment,
* can do PGE,
* do not have a hearing problem or a communication disability will be admitted.

Exclusion Criteria:

* who were discharged early,
* had an unexpected change in their condition,
* started to experience pain,
* could not adapt to the working principles,
* gave up volunteering will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-05-09 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
sleep quality, | 06.00 am the day before the progressive relaxation exercise
  Richard's Campbell Sleep Scale (RCS) consists of 6 items. In the scale, patients are asked to evaluate between 0 and 100 points for each item. The 6th item, which evaluates the noise level in the environment, is not included in the total score evaluation. The result is obtained by dividing the total score obtained from the scale by the number of questions, and "0-25" points indicate "very bad sleep" and "76-100" points indicate "very good sleep".
melatonin and serotonin in urine | 06.00 am the day before the progressive relaxation exercise
  In order to determine the levels of serotonin metabolite 5-hydroxyindolacetic acid (5-HIAA) and melatonin metabolite 6-sulphatoxymelatonin from patients in the experimental and control groups, urine samples will be taken between 23:00 at night and 07:00 in the morning at the end of the first and fourth day. On the 5th day, after the last urine taken in the morning is added, a urine sample will be taken into a sample container containing 10-15 ml of 6 M HCl and stored at -80 degrees for analysis in the biochemistry laboratory.

SECONDARY OUTCOMES:
sleep quality, | 06.00 am, after 3 consecutive days of progressive relaxation exercise
  Richard's Campbell Sleep Scale (RCS) consists of 6 items. In the scale, patients are asked to evaluate between 0 and 100 points for each item. The 6th item, which evaluates the noise level in the environment, is not included in the total score evaluation. The result is obtained by dividing the total score obtained from the scale by the number of questions, and "0-25" points indicate "very bad sleep" and "76-100" points indicate "very good sleep".
melatonin and serotonin in urine | 06.00 am the day after the progressive relaxation exercise
  In order to determine the levels of serotonin metabolite 5-hydroxyindolacetic acid (5-HIAA) and melatonin metabolite 6-sulphatoxymelatonin from patients in the experimental and control groups, urine samples will be taken between 23:00 at night and 07:00 in the morning at the end of the first and fourth day. On the 5th day, after the last urine taken in the morning is added, a urine sample will be taken into a sample container containing 10-15 ml of 6 M HCl and stored at -80 degrees for analysis in the biochemistry laboratory.

CONTACTS AND LOCATIONS:
Overall Officials: Tunç ELİŞ, Principal Investigator — Kafkas Universıty/Turkey
Locations (2):
- Turkey (Türkiye) (2):
  - Atatürk University, Erzurum
  - Ataturk Üniversity, Erzurum

IPD SHARING:
Plan to Share IPD: No